CLINICAL TRIAL: NCT03292809
Title: A Phase 2b/3, Multicenter, Randomized, Double-masked, Vehicle-controlled Clinical Study to Assess the Efficacy and Safety of Topical CyclASol® for the Treatment of Signs and Symptoms of Dry Eye Disease (DED) (ESSENCE Trial)
Brief Title: CyclASol for the Treatment of Signs and Symptoms of Dry Eye Disease (DED)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYS-003 (ESSENCE)
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions; Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CyclASol Ophthalmic Solution (Experimental): Cylclosporine A solution in vehicle
  Interventions: Drug: CyclASol topical ocular, eye drops
- Vehicle Ophthalmic Solution (Placebo Comparator): Vehicle only
  Interventions: Drug: Vehicle topical ocular, eye drops

INTERVENTIONS:
Drug: CyclASol topical ocular, eye drops — Cyclosporine A solution in vehicle
  Other Names: Ciclosporine (CsA)
  Arms: CyclASol Ophthalmic Solution
Drug: Vehicle topical ocular, eye drops — Vehicle
  Other Names: Vehicle
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
The objective of this study is to assess the efficacy, safety, and tolerability of CyclASol Ophthalmic Solution in comparison to vehicle for the treatment of the signs and symptoms of DED.

DETAILED DESCRIPTION:
This Phase 2b/3 study will assess the efficacy, safety and and tolerability of CyclASol Ophthalmic Solution as one drop twice daily versus vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF (Informed Consent Form) and HIPAA (Health Insurance Portability and Accountability Act)
* Patient-reported history of DED in both eyes
* Current use of OTC (over-the-counter) and/or artificial tears for dry eye symptoms
* Ability and willingness to follow instructions, including participation in all study assessments and visits

Exclusion Criteria:

* Women who are pregnant, nursing or planning a pregnancy
* Unwillingness to submit a urine pregnancy test at screening and the last visit (or early termination visit) if of childbearing potential, or unwillingness to use acceptable means of birth control
* Clinically significant slit-lamp findings or abnormal lid anatomy at screening
* Ocular/periocular malignancy
* History of herpetic keratitis
* Active ocular allergies or ocular allergies that may become active during the study period
* Ongoing ocular or systemic infection at screening or baseline
* Wear of contact lenses within 3 months prior to screening or anticipated use of contact lenses during the study
* History of no response to previous topical Cyclosporine A and/or use of topical Cyclosporine A or Liftigrast within 2 months prior to screening
* Intraocular surgery or ocular laser surgery within the previous 6 months, or have any planned ocular and/or lid surgeries over the study period
* Presence of uncontrolled systemic diseases
* Presence of known allergy and/or sensitivity to the study drug or its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Kroesser, PhD, Study Director — Novaliq GmbH
Locations (9):
- United States (9):
  - CYS-003 Investigational Site, Newport Beach, California
  - CYS-003 Investigational Site, Torrance, California
  - CYS-003 Investigational Site, Indianapolis, Indiana
  - CYS-003 Investigational Site, Louisville, Kentucky
  - CYS-003 Investigational Site, Andover, Massachusetts
  - CYS-003 Investigational Site, Raynham, Massachusetts
  - CYS-003 Investigational Site, Memphis, Tennessee
  - CYS-003 Investigational Site, Nashville, Tennessee
  - CYS-003 Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sheppard JD, Wirta DL, McLaurin E, Boehmer BE, Ciolino JB, Meides AS, Schluter T, Ousler GW, Usner D, Krosser S. A Water-free 0.1% Cyclosporine A Solution for Treatment of Dry Eye Disease: Results of the Randomized Phase 2B/3 ESSENCE Study. Cornea. 2021 Oct 1;40(10):1290-1297. doi: 10.1097/ICO.0000000000002633. PMID 34481407
- [Derived] Akpek EK, Sheppard JD, Hamm A, Angstmann-Mehr S, Krosser S. Efficacy of a new water-free topical cyclosporine 0.1% solution for optimizing the ocular surface in patients with dry eye and cataract. J Cataract Refract Surg. 2024 Jun 1;50(6):644-650. doi: 10.1097/j.jcrs.0000000000001423. PMID 38334413
- See also: Publication of Study Results — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8423142/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After a 2-week run-in period, eligible DED patients were randomized 1:1 to either CyclASol 0.1% or vehicle twice daily.
Period: Overall Study
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Started | 162 | 166
Completed | 155 | 163
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution | Total
Number analyzed (Participants) | 162 | 166 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (13.6) | 61.3 (12.66) | 61.4 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 119 | 235
  Male | 46 | 47 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 11 | 26
  Not Hispanic or Latino | 147 | 155 | 302
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 14 | 19 | 33
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 16 | 14 | 30
  White | 130 | 127 | 257
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 162 | 166 | 328

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Corneal Fluorescein Staining at Day 29
Description: CFS was assessed in each eye using the National Eye Institute (NEI) scale.
  A standardized grading system of 0-3 is used for each of the five areas on each cornea. Grade 0 will be specified when no staining is present. The maximum total score for each eye is 15. Higher values describe greater staining and corneal damage.
Time Frame: baseline and 1 month [day 29]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 162 | 166
score on a scale | -2.9 (2.59) | -2.2 (2.73)

2. Primary Outcome: Change From Baseline in Ocular Surface Disease Index at Day 29
Description: The OSDI score is a composite measure built on 12 questions,with totals ranging from 0 to 100, and higher scores representing a worse disease index.
Time Frame: baseline and 1 month [day 29]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 162 | 166
score on a scale | -7.08 (18.650) | -5.37 (15.291)

ADVERSE EVENTS:
Time Frame: 85 Days ± 2 (Randomization until Study Exit)
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/166
Serious Adverse Events (participants affected / at risk) | 0/162 | 3/166
Other Adverse Events (participants affected / at risk) | 26/162 | 23/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CyclASol Ophthalmic Solution (N=162) | Vehicle Ophthalmic Solution (N=166)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Degenerated disc disease L1-L4
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CyclASol Ophthalmic Solution (N=162) | Vehicle Ophthalmic Solution (N=166)
Visual acuity reduced (Eye disorders) | 5 | 3
Instillation site pain (Eye disorders) | 4 | 2
Vision blurred (Eye disorders) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 8 | 7
Nasopharyngitis (Infections and infestations) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT03292809/Prot_SAP_000.pdf